CLINICAL TRIAL: NCT05160753
Title: Laparoscopic Gastric Function Preserving Surgery Combined With Resection of the Anterior Lymphatic Drainage Area. Comparison of Laparoscopic Standard Radical Gastric Cancer Surgery for Early Distal Gastric Cancer Multicenter, Prospective, Randomized, Open, Parallel-controlled, Non-inferiority Efficacy Clinical Trial
Brief Title: Laparoscopic Gastric Function Preserving Surgery Combined With Resection of the Anterior Lymphatic Drainage Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Tongzhou District Hospital (Unknown); Haimen People's Hospital (Unknown); Dongtai People's Hospital (Unknown); Qidong City People's Hospital (Unknown); Rudong County Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Qinsheng Mao, professor, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LGFPS
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-02

CONDITIONS: Gastric Cancer Stage I
Keywords: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: 1. The group of laparoscopic gastric function preserving surgery combined with resection of the anterior lymphatic drainage area.
  2. Patients in the control group will undergo standard laparoscopic gastrectomy (laparoscopic distal gastrectomy with simultaneous D1+ lymph node dissection).
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gastric function preserving surgery combined with resection of the anterior lymphatic drainage area. (Experimental): 1. Steps of sentinel lymph node dissection Indocyanine green (ICG) tracing of anterior lymph nodes. ICG injection: A 4mL volume of double tracer is injected into the submucosa of the four quadrants of the primary tumor by intraoperative gastroscopic method. 0.5 mL was injected at each site, and 15 minutes after gastroscopic tracer injection, the green anterior lymph nodes were carefully dissected and removed from the surgical area and evaluated for lymph node metastasis by parallel intraoperative freezing.
  2. Intraoperative and postoperative pathological examination Intraoperative histological examination of lymph nodes collected from the anterior lymph node pool was performed, If all collected anterior lymph nodes are negative, laparoscopic gastric function preserving surgery will be performed. After surgery, anterior lymph nodes that proved to be tumor-free on intraoperative frozen section examination were reevaluated.
  Interventions: Procedure: Laparoscopic gastric function preserving surgery combined with resection of the anterior lymphatic drainage area
- Patients in the control group will undergo standard laparoscopic gastrectomy (Active Comparator): Patients in the control group will undergo standard laparoscopic gastrectomy (laparoscopic distal gastrectomy with simultaneous D1+ lymph node dissection).
  Interventions: Procedure: Laparoscopic gastric function preserving surgery combined with resection of the anterior lymphatic drainage area

INTERVENTIONS:
Procedure: Laparoscopic gastric function preserving surgery combined with resection of the anterior lymphatic drainage area — A 4mL volume of double tracer is injected into the submucosa of the four quadrants of the primary tumor by intraoperative gastroscopic method., and 15 minutes after gastroscopic tracer injection, the green anterior lymph nodes were carefully dissected and removed from the surgical area and evaluated for lymph node metastasis by parallel intraoperative freezing.If all collected anterior lymph nodes are negative, laparoscopic gastric function preserving surgery will be performed.

SUMMARY:
Nowadays, while pursuing the eradication of tumor, how to maximize the preservation of normal anatomy and physiological functions of the stomach, reduce the surgical trauma caused by excessive debridement, and improve the quality of life of patients after surgery has become a more important concern in the treatment of early gastric cancer. This prospective multicenter randomized controlled clinical trial was designed to elucidate the oncologic safety of laparoscopic gastric preservation surgery compared to standard laparoscopic gastrectomy. The oncologic safety of laparoscopic gastric preservation surgery with anterior basal dissection (SBD) compared to standard laparoscopic gastrectomy. This trial is an investigator-initiated, multicenter, prospective, randomized, open, parallel-controlled with a non-inferiority design. Patients diagnosed as distal gastric cancer with clinical stage T1N0M0, with a lesion diameter of 3 cm or less were eligible to participate in this study. Patients will be randomized to either laparoscopic stomach-preserving surgery with SBD or standard surgery. The primary end-point is 3-year disease-free survival.

ELIGIBILITY:
Inclusion Criteria：

1. single lesion detected by gastroscopy and clearly diagnosed histologically as gastric adenocarcinoma.
2. patients with gastric cancer with clinical stage T1N0M0 (based on the TNM stage of the 8th edition of AJCC) (T-stage assessed by ultrasound gastroscopy and N-stage and M-stage assessed by enhanced CT).
3. tumor length diameter less than 3 cm.
4. the lesion is located in the gastric sinus.
5. patient age greater than 20 years and less than 80 years.
6. ECOG score of 0 or 1.
7. The patient voluntarily participated in this clinical study.

Exclusion Criteria:

1. Patients with gastric cancer suitable for endoscopic treatment (differentiated gastric cancer with tumor length diameter less than 2 cm and located within the mucosa).
2. cardiopulmonary dysfunction that cannot tolerate laparotomy.
3. pyloric duct gastric cancer.
4. Previously undergone upper abdominal surgery.
5. other malignant tumors diagnosed within the previous five years.
6. Pregnant women.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) at three years | three years
  The criteria for DFS events in this study were as follows: recurrence of the primary tumor at the incisional margin or anastomosis, heterochronic metastasis in the remnant stomach, histologically or imaging confirmed intraperitoneal recurrence, lymph node metastasis, distant metastasis, new malignancy in other organs, and other causes of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miwa K, Kinami S, Taniguchi K, Fushida S, Fujimura T, Nonomura A. Mapping sentinel nodes in patients with early-stage gastric carcinoma. Br J Surg. 2003 Feb;90(2):178-82. doi: 10.1002/bjs.4031. PMID 12555293
- [Background] Kitagawa Y, Takeuchi H, Takagi Y, Natsugoe S, Terashima M, Murakami N, Fujimura T, Tsujimoto H, Hayashi H, Yoshimizu N, Takagane A, Mohri Y, Nabeshima K, Uenosono Y, Kinami S, Sakamoto J, Morita S, Aikou T, Miwa K, Kitajima M. Sentinel node mapping for gastric cancer: a prospective multicenter trial in Japan. J Clin Oncol. 2013 Oct 10;31(29):3704-10. doi: 10.1200/JCO.2013.50.3789. Epub 2013 Sep 9. PMID 24019550
- [Background] Lips DJ, Schutte HW, van der Linden RL, Dassen AE, Voogd AC, Bosscha K. Sentinel lymph node biopsy to direct treatment in gastric cancer. A systematic review of the literature. Eur J Surg Oncol. 2011 Aug;37(8):655-61. doi: 10.1016/j.ejso.2011.05.001. Epub 2011 Jun 1. PMID 21636243
- [Background] Takahashi N, Nimura H, Fujita T, Mitsumori N, Shiraishi N, Kitano S, Satodate H, Yanaga K. Laparoscopic sentinel node navigation surgery for early gastric cancer: a prospective multicenter trial. Langenbecks Arch Surg. 2017 Feb;402(1):27-32. doi: 10.1007/s00423-016-1540-y. Epub 2016 Dec 20. PMID 27999935